CLINICAL TRIAL: NCT03712878
Title: A 2 Step Approach to Matched Related Hematopoietic Stem Cell Transplantation for Patients With Hematological Malignancies-5+5 Dosing
Brief Title: 2-Step Approach to Stem Cell Transplant in Treating Participants With Hematological Malignancies
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sidney Kimmel Cancer Center at Thomas Jefferson University (Other)
Responsible Party: Sponsor
Organization: Thomas Jefferson University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 18D.419; JT 12822 (Other: JeffTrial Number)
Record Dates: First submitted 2018-10-17; First posted 2018-10-19 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Hematopoietic and Lymphoid Cell Neoplasm
MeSH Terms: conditions — Hematologic Neoplasms | interventions — Whole-Body Irradiation; Cyclophosphamide; Stem Cell Transplantation; Tacrolimus; Mycophenolic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Treatment (TBI, DLI, chemotherapy, HSCT, tacrolimus, MMF) (Experimental): Description CONDITIONING REGIMEN: Participants undergo TBI BID on days -9 to -6.
  TRANSPLANT: Participants receive donor lymphocytes IV on day -6 after the last dose of TBI.
  CONDITIONING REGIMEN: Participants receive cyclophosphamide IV on days -3 and -2.
  TRANSPLANT: Participants undergo hematopoietic stem cell transplantation on day 0.
  GVHD PROPHYLAXIS: Participants receive tacrolimus IV beginning on day -1 with taper beginning on day 42 in the absence of GVHD, a suspicion of GVHD, or previous history of GVHD requiring a taper delay. Participants also receive mycophenolate mofetil IV BID beginning on day -1 through day 28 in the absence of GVHD.
  Interventions: Radiation: Total-Body Irradiation; Procedure: Donor Lymphocyte Infusion; Drug: Cyclophosphamide; Procedure: Allogeneic Hematopoietic Stem Cell Transplantation; Drug: Tacrolimus; Drug: Mycophenolate Mofetil

INTERVENTIONS:
Radiation: Total-Body Irradiation — Undergo TBI
  Other Names: SCT_TBI; TBI; TOTAL BODY IRRADIATION; Whole Body; Whole Body Irradiation; Whole-Body Irradiation
Procedure: Donor Lymphocyte Infusion — Given IV
  Other Names: DLI; Donor Leukocyte Infusion
Drug: Cyclophosphamide — Given IV
  Other Names: (-)-Cyclophosphamide; 1-bis(2-chloroethyl)-amino-1-oxo-2-aza-5-oxaphosphoridin monohydrate; 2-[bis(2-chloroethyl)amino]tetrahydro-2H-1,3,2-oxazaphosphorine 2-oxide monohydrate; 2-[bis(b-chloroethyl)amino]-1-oxa-3-aza-2-phosphacyclohexane-2-oxide monohydrate; 2-[di(chloroethyl)amino]-1-oxa-3-aza-2-phosphacyclohexane 2-oxide monohydrate; 2H-1,3,2-Oxazaphosphorine; 2-[bis(2-chloroethyl)amino]tetrahydro; 2-oxide, monohydrate; 6055-19-2; bis(2-chloroethyl)phosphamide cyclic propanolamide ester monohydrate; Bis(2-chloroethyl)phosphoramide cyclic propanolamide ester monohydrate; Carloxan; Ciclofosfamida; Ciclofosfamide; Cicloxal; Clafen; Claphene; CP monohydrate; CTX; CYCLO-cell; Cycloblastin; Cycloblastine; Cyclophospham; Cyclophosphamid monohydrate; Cyclophosphamide Monohydrate; Cyclophosphamidum; Cyclophosphan; Cyclophosphane; Cyclophosphanum; Cyclostin; Cyclostine; Cytophosphan; Cytophosphane; Cytoxan; Fosfaseron; Genoxal; Genuxal; Ledoxina; Mitoxan; N,N-bis(2-chloroethyl)-N',O-propylenephosphoric acid ester diamide monohydrate; N,N-bis(2-chloroethyl)-N'-(3-hydroxypropyl)phosphorodiamidic acid intramolecular ester monohydrate; N,N-bis(2-chloroethyl)tetrahydro-2H-1,3,2-oxazaphosphorin-2-amine 2-oxide monohydrate; N,N-bis(b-chloroethyl)-N',O-trimethylenephosphoric acid ester diamide monohydrate; N,N-bis(beta-chloroethyl)-N',O-propylenephosphoric acid ester diamide monohydrate; N,N-bis(beta-chloroethyl)-N',O-trimethylenephosphoric acid ester diamide monohydrate; Neosar; Revimmune; Syklofosfamid; WR- 138719
Procedure: Allogeneic Hematopoietic Stem Cell Transplantation — Undergo HSCT
  Other Names: Allogeneic; Allogeneic Hematopoietic Cell Transplantation; allogeneic stem cell transplantation; HSC; HSCT; Stem Cell Transplantation
Drug: Tacrolimus — Given IV
  Other Names: 109581-93-3; FK 506; Fujimycin; Hecoria; Prograf; Protopic
Drug: Mycophenolate Mofetil — Given IV
  Other Names: 115007-34-6; 128794-94-5; Cellcept; MMF

SUMMARY:
This phase II trial studies how well a 2-step approach to stem cell transplant works in treating patients with blood cancers. Giving chemotherapy and total body irradiation before a lymphocyte (white blood cell) and stem cell transplant helps stop the growth of cells in the bone marrow including normal blood-forming cells (stem cells) and cancer cells. By giving the donor cells in two steps, the dose of lymphocytes given can be tightly controlled and they can be made more tolerant to the body. When the healthy lymphocytes and stem cells from a donor are infused into the patient, they may help the patient's bone marrow make stem cells, red blood cells, white blood cells, and platelets. Sometimes the transplanted cells from a donor can make an immune response against the body's normal cells called graft versus host disease. Giving tacrolimus and mycophenolate mofetil may stop this from happening.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess whether providing a patient with "5+5" dosing in a 2 step matched related donor hematopoietic stem cell transplantation (HSCT) increases the percentage of patients who achieve full donor chimerism earlier as defined by 98% or greater donor T cell chimerism at 28 days post HSCT (d+28).

SECONDARY OBJECTIVES:

I. To assess day (d) +90 chimerism in patients receiving "5+5" dosing. II. To assess post HSCT relapse rates in patients receiving "5+5" dosing. III. To assess rates of grade II-IV graft versus host disease (GVHD) in patients receiving "5+5" dosing.

IV. To assess treatment-related mortality (TRM) in patients receiving "5+5" dosing.

EXPLORATORY OBJECTIVES:

I. To assess whether patients receiving "5+5" dosing have lower rates of cytomegalovirus (CMV) reactivation as compared to patients treated on Thomas Jefferson University (TJU) 08D.85 (1st Generation 2-Step Matched Related Trial).

OUTLINE:

CONDITIONING REGIMEN: Patients undergo total body irradiation (TBI) twice daily (BID) on days -9 to -6.

TRANSPLANT: Patients receive donor lymphocytes intravenously (IV) on day -6 after the last dose of TBI.

CONDITIONING REGIMEN: Patients receive cyclophosphamide IV on days -3 and -2.

TRANSPLANT: Patients undergo hematopoietic stem cell transplantation on day 0.

GVHD PROPHYLAXIS: Patients receive tacrolimus IV beginning on day -1 with taper beginning on day 42 in the absence of GVHD, a suspicion of GVHD, or previous history of GVHD requiring a taper delay. Patients also receive mycophenolate mofetil IV BID beginning on day -1 through day 28 in the absence of GVHD.

After completion of study treatment, patients are followed up at days 28, 90, 180, 270, and 365.

ELIGIBILITY:
Inclusion Criteria:

* Provide signed and dated informed consent form.
* Have a hematological malignancy or any type of dyscrasia in which allogeneic HSCT is thought to be beneficial.
* Have a related donor who is no more than a 1-antigen mismatch at the human leukocyte antigen (HLA)-A; B; C; DR loci in the GVHD direction with the patient. (Patients with a syngeneic donor may be treated on this therapeutic approach, but their outcomes will not be part of the statistical aims of the study.
* LVEF (left ventricular end diastolic function) of >= 45%.
* DLCO (diffusing capacity of the lung for carbon monoxide) >= 50% of predicted corrected for hemoglobin.
* FEV-1 (forced expiratory volume at 1 second >= 50% of predicted.
* Serum bilirubin =< 1.8.
* Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) =< 2.5 x upper limit of normal.
* Creatinine clearance of >= 60 mL/min.
* Have a Hematopoietic Cell Transplant Comorbidity Index (HCT-CI) score =< 5 points (patients with greater than 5 points will be allowed for trial with approval of the principal investigator [PI] and at least 1 co-investigator [co-I] not on the primary care team of the patient). This is an adjustment to account for healthy patients who meet the spirit of this protocol but have histories that result in higher than HCT-CI 5 points. An example is a patient with a solid tumor malignancy in their remote history (adds 3 points to HCT-CI total) where the treatment for the malignancy occurred years to decades before and there has been complete recovery of toxicities.
* Have a Karnofsky performance score (KPS) >= 80%.
* Women of reproductive potential (defined as women under the age of 50 years still menstruating within 2 months of HSCT despite past history of chemotherapy) will be counseled to use highly effective contraception including oral, intramuscular (IM), or patch contraceptives, intrauterine device (IUD), diaphragm, cervical cap, or contraceptive implant. Pharmacological avoidance of pregnancy and suppression of menstruation may be instituted during the HSCT inpatient stay.
* Men will be asked to abstain from sexual relations during the treatment period of the HSCT stay.
* DONOR: All donors are selected and screened for their ability to provide adequate infection-free apheresis products for the patient in a manner that does not put the donor at risk for negative consequences.

Exclusion Criteria:

* Be human immunodeficiency virus (HIV) positive.
* Be pregnant or breastfeeding.
* Have received alemtuzumab or rabbit antithymocyte globulin (ATG) within 8 weeks or horse ATG within 6 weeks of the transplant admission. This exclusion criterion will be documented by the absence of these drugs in the medical record.
* Patients with evidence of another malignancy, exclusive of a skin cancer that requires only local treatment, should not be enrolled on this protocol without the specific approval of the PI. If the PI disregards this criterion (example of this is localized prostate cancer not yet requiring treatment), the rationale must be documented in the study binder). This exclusion criterion will be documented by the absence of these drugs in the medical record.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2018-09-19 (Actual); Primary Completion 2025-03-19 (Actual); Study Completion 2025-03-19 (Actual)

PRIMARY OUTCOMES:
Donor T cell chimerism | At day +28
  For chimerism rates, the method of Atkinson and Brown will be used to allow for the two-stage design. Will be presented with corresponding 95% confidence intervals.

SECONDARY OUTCOMES:
Donor T cell chimerism | At day +90
  Will be presented with corresponding 95% confidence intervals. For chimerism rates, the method of Atkinson and Brown will be used to allow for the two-stage design.
Relapse rate | At 1 year post-hematopoietic stem cell transplantation (HSCT)
  Will be presented with corresponding 95% confidence intervals.
Incidence of grades II-IV graft versus host disease (GVHD) | Within 1 year of HSCT
  Will be presented with corresponding 95% confidence intervals.
Rate of treatment-related mortality (TRM) | At 1 year post-HSCT
  Will be presented with corresponding 95% confidence intervals.

OTHER OUTCOMES:
Rate of cytomegalovirus | Up to 100 days
  Rate of cytomegalovirus

CONTACTS AND LOCATIONS:
Overall Officials: USAMA GERGIS, MD, Principal Investigator — Sidney Kimmel Cancer Center at Thomas Jefferson University
Locations (1):
- Sidney Kimmel Cancer Center at Thomas Jefferson University, Philadelphia, Pennsylvania, United States

REFERENCES:
- See also: Thomas Jefferson University Hospital — http://hospitals.jefferson.edu/